CLINICAL TRIAL: NCT06356740
Title: Randomized Pilot Trial to Evaluate the Efficacy and Tolerance of Abacavir/Lamivudine Treatment in Patients With Systemic Lupus Erythematosus (PENCIL)
Brief Title: Efficacy and Tolerance of Abacavir/Lamivudine Treatment in Patients With Systemic Lupus Erythematosus
Acronym: PENCIL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL22_0878; 2023-508611-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus; Systemic Lupus Erythematosus; abacavir; lamivudine; nucleoside reverse transcriptase inhibitors
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection; Lamivudine

STUDY DESIGN:
Intervention Model Description: Open-label randomized, controlled study with 2 parallel arms (Add-on treatment versus standard of care treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abacavir 600 mg/lamivudine 300 mg (Experimental): Patients randomized to this group will take 1 tablet (600 mg lamivudine and 300 mg abacavir) once daily for 6 months in addition to their usual treatment.
  Interventions: Biological: Blood sample; Drug: Treatment :Abacavir 600 mg/lamivudine 300 mg; Other: Lupus Impact Tracker questionnaire
- Control group (standard of care) (Active Comparator): Patients randomized to this group will continue their usual treatment for lupus systemic.
  Interventions: Biological: Blood sample; Other: Lupus Impact Tracker questionnaire

INTERVENTIONS:
Biological: Blood sample — blood test to assess :
  * human leukocyte antigen (HLA)-B*5701 status to identify risk of allergy or hypersensitivity to abacavir (the study treatment)
  * IFN-signature ans IFN-alpha dosage
  * human immunodeficiency virus (HIV), hepatitis B virus (HBV) and Hepatitis C virus (HCV) serologies
  * Human chorionic gonadotropin (βHCG)
  * HERVs dosage A biological collection will also be created. The total volume of blood collected specifically for the research for the entire duration of the study is 62.5 millilitre (mL) maximum.
Drug: Treatment :Abacavir 600 mg/lamivudine 300 mg — Patients randomised to the experimental arm will be required to take 1 tablet (600 mg lamivudine and 300 mg abacavir) once daily for 6 months in addition to their usual treatment.
  Arms: Abacavir 600 mg/lamivudine 300 mg
Other: Lupus Impact Tracker questionnaire — Patients will be asked to complete the Lupus Impact Tracker questionnaire at visit V1 (randomisation visit), visit 3 (at 6 months of treatment) and visit 4 (12 months after visit 1).

SUMMARY:
Systemic lupus (SL) is a rare chronic autoimmune disease characterized by the production of autoantibodies directed against nuclear antigens, particularly native double-stranded deoxyribonucleic acid (DNA), and excessive production of antiviral cytokines: type I interferons, particularly interferon alpha (IFN-α). IFN-α production results from the excessive detection of nucleic acids (DNA or Ribonucleic Acid (RNA)) by endosomal or intracytoplasmic receptors that are capable of inducing interferon production. The precise mechanisms of cytoplasmic sensor activation remain unknown; however, recent work in the field of interferonopathies suggests a role for human endogenous retroviruses (HERVs). HERVs are remnants of ancient infections caused by exogenous retroviruses integrated into the genome during evolution and represent 8% of the human genome.Several studies have suggested a role for HERVs in the development and maintenance of an excessive immune response in lupus patients and other autoimmune diseases by affecting the type I interferons (I IFN) signalling pathway.

To date, none of the approved immunosuppressive drugs for Systemic Lupus Erythematosus (SLE) have been shown to be effective in the background treatment of SL or in preventing relapse. Consequently, there is an urgent need to identify new molecules and therapeutic avenues for disease-modifying therapies.

In this study, an innovative therapeutic strategy using a combination of nucleoside reverse transcriptase inhibitors (NRTIs), abacavir/lamivudine, is proposed to treat SLE. Thus, we propose a pilot Phase II, randomized, open-label study using NRTIs in patients with SL in remission or with low clinical activity, and evaluating a biological endpoint (IFN signature), which is a direct proxy for the drug's expected effect.

The main objective is to compare the addition of Abacavir/Lamivudine (Add-on) to standard care for 6 months, on the value of the interferon (IFN) transcriptomic signature of patients with systemic lupus with low activity as defined by the Lupus Low Disease Activity State (LLDAS).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥12 years old (weighing more than 25 kg) and ≤ 65 years old
* Diagnosis of SL according to 2019 American College of rheumatology (ACR) / European Ligue against Rheumatism (EULAR) criteria (score >10)
* Patient with SL in remission or with low clinical activity according to LLDAS disease criteria
* For patients (including sexually active adolescents) of childbearing age, effective contraception (sexual abstinence, hormonal contraception, intrauterine device or hormone-releasing system, cap, diaphragm, sponge with spermicide, or condom) for the entire duration of treatment is required. Pregnancy tests will be performed according to the inclusion criteria.
* Patient affiliated to a social security scheme
* Free, informed and written consent signed by patient or parents/legal guardian

Exclusion Criteria:

* Patients with HLA-B*5701 status (risk of allergy or hypersensitivity to Abacavir)
* History of allergy or hypersensitivity to abacavir, lamivudine, or excipients (tablet core: microcrystalline cellulose, crospovidone, magnesium stearate, colloidal anhydrous silica, talc; film coating: hypromellose, titanium dioxide (E171), macrogol, polysorbate 80).
* Patients on anti-retroviral therapy
* Patients with chronic HIV, HBV or HCV infection
* Pregnant or breast-feeding woman
* Patient treated with Lamivudine and/or Abacavir
* Patient treated with a cytidine analog
* Patient on treatment containing Cladribine
* Patient on treatment containing a trimethoprim/sulfamethoxazole combination
* Patients with renal insufficiency (creatinine clearance < 50 ml/min)
* Patients with moderate or severe hepatic impairment (prothrombin level <50%)
* Patient participating in other interventional drug research

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Absolute variation in interferon signature (IFN) | At M6 (after 6 months of treatment)
  Absolute change in interferon (IFN) signature will be assessed between the start of treatment (M0) and after 6 months of treatment (M6) in the total population (then in the pediatric population, then in the adult population)..

SECONDARY OUTCOMES:
percentage of patients maintaining LLDAS criteria | until 12 months after randomisation
  The percentage of patients maintaining LLDAS criteria will be assessed at M6 and M12 in the 2 arms.
number of relapses | until 12 months after randomisation
  number of relapses and time to relapse between M0 and M12 (collected continuously) will be assessed
anti-native double-stranded DNA quantification | until 12 months after randomisation
  Evaluation of the effect of treatment on lupus biomarkers by quantifying anti-native double-stranded DNA
anti-extractable nuclear antigens (anti-ENA) quantification | until 12 months after randomisation
  Evaluation of the effect of treatment on lupus biomarkers by quantifying anti-ENA
interferon-α production quantification | until 12 months after randomisation
  Evaluation of the effect of treatment on lupus biomarkers by interferon-α production
Number of successful patients | until 6 months after randomisation
  The number of patients in each arm achieving success will be assessed. Success is defined as a ≥50% reduction in IFN signature between M0 and M6.
Cumulative dose of intravenous (IV) corticosteroids | until 12 months after randomisation
  The impact of treatment on corticosteroid intake in the "Intervention" arm and the "No intervention" arm at M control arm will be assessed by observing the cumulative dose of intravenous (IV) and oral corticosteroids.
Lupus Impact Tracker questionnaire score | until 12 months after randomisation
  Quality of life will be assessed by comparing Lupus Impact Tracker™ questionnaire scores at M6 and M12 in the Intervention arm and control arm.
  The lupus impact tracker (LIT) is a 10-item patient reported outcome tool to measure the impact of systemic lupus erythematosus or its treatment on patients' daily lives. Each answer is marked from 0 to 4 points. The lower the Lupus Impact score, the less impact lupus is having on the life of patient.
number of missed treatment | until 6 months after randomisation
  Adherence to treatment will be assessed by recording the number of doses missed and the reasons for missed doses.
number of adverse event (AE) | until 12 months after randomisation
  To assess the safety and tolerability of the drug, the number of AE will be compared between the two randomisation arms.
number of serious adverse event (SAE) | until 12 months after randomisation
  To assess the safety and tolerability of the drug, the number of SAE will be compared between the two randomisation arms.
HERVs transcription quantification | until 12 months after randomisation
  The difference in HERVs copy number in the 2 arms will be assessed. A comparison between groups will be performed.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Groupe Hospitalier Pellegrin-CHU de Bordeaux, Bordeaux
  - Hôpital Femme-Mère-Enfant (HCL), Bron
  - CHU de Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Nord de Grenoble - Albert Michallon, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital de la Croix-Rousse (HCL), Lyon
  - Hôpital Edouard Herriot (HCL), Lyon
  - Hôpital Necker-Enfants malades, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Lyon Sud (HCL), Pierre-Bénite
  - CHU de Saint-Etienne - Hôpital Nord, Saint-Priest-en-Jarez